CLINICAL TRIAL: NCT05261919
Title: Meridian Study on the Response Current Affected by Acupuncture Needling Direction
Brief Title: Relationship Between Acupuncture Needling Direction and Electric Current
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201901601A3
Record Dates: First submitted 2022-02-14; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2020-01

CONDITIONS: Acupuncture; Electricity; Effects
Keywords: Acupuncture; Directional manipulation; Electricity; Meridian theory; Traditional Chinese medicine; Supplementation; Draining

STUDY DESIGN:
Intervention Model Description: All the participants were in one group and received acupuncture manipulation. The investigator used directional supplementation and draining manipulation. The investigator perform acupuncture with supplementation manipulation first, followed by a measurement of the electrical characteristics using Agilent B1500A. The investigator remove the acupuncture and then perform acupuncture with draining manipulation, followed by measurements. After one meridian measurements were completed, the investigator removed the needle and proceeded to the next meridian to repeat the same procedure.
  The supplementation manipulation is defined as the angle of needle insertion to skin as 45 degrees with the needle tip in the same direction as the meridian. While the draining manipulation is defined as the angle of needle insertion at 45 degrees with the needle tip direction opposite to that of the meridian.
  The acupoints were HT7、HT3、SI5、SI8、BL57、BL40、KI3、KI10 in this study.
Masking Description: There were no masking in this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- acupuncture with manipulation group (Experimental): 30 participant were recruited in this study. All the participants received acupuncture at the acupoints (HT7、HT3、SI5、SI8、BL57、BL40、KI3、KI10) and were measured by an Agilent B1500A semiconductor analyzer.
  The investigator perform acupuncture with supplementation manipulation first, followed by a measurement of the electrical characteristics using Agilent B1500A. The investigator remove the acupuncture and then perform acupuncture with draining manipulation, followed by measurements. After one meridian measurements were completed, the investigator removed the needle and proceeded to the next meridian to repeat the same procedure.
  Interventions: Procedure: Acupuncture manipulation

INTERVENTIONS:
Procedure: Acupuncture manipulation — The investigator used directional supplementation and draining manipulation. The supplementation manipulation is defined as the angle of needle insertion to skin as 45 degrees with the needle tip in the same direction as the meridian. While the draining manipulation is defined as the angle of needle insertion at 45 degrees with the needle tip direction opposite to that of the meridian.
  Other Names: Directional manipulation

SUMMARY:
This study applies a semiconductor analyzer to investigate the effects of acupuncture manipulation.

DETAILED DESCRIPTION:
Acupuncture manipulation with needling direction is important for the therapeutic effect based on traditional Chinese medicine theory. However, research usually focuses on the therapeutic effects on the acupoints and acupuncture time rather than on the manipulation method. This study applies a semiconductor analyzer to investigate the effects of acupuncture manipulation.

30 healthy participants were recruited in the study. This study employed an Agilent B1500A semiconductor analyzer to investigate the electric characteristics of meridians under directional supplementation and draining manipulation. We measured the electric current of meridians under different manipulation, and compared the difference between supplementation and draining manipulation in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* at least 20 years old
* agree to the informed consent

Exclusion Criteria:

* under 20 years old
* pregnant or breast-feeding women
* those with an empty stomach before the study
* a tendency toward bleeding with thrombocytopenia or history of platelets < 20000 or a user of an anti-platelet drug.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
The electric current | through study completion, an average of 90 minutes
  Agilent B1500A is a device that can measure the electric current after acupuncture manipulation. The investigators measure the electric current after intervention of supplementation manipulation and draining manipulation respectively.
The voltage | through study completion, an average of 90 minutes
  Agilent B1500A is a device that can measure the voltage after acupuncture manipulation. The investigators measure the voltage after intervention of supplementation manipulation and draining manipulation respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chiang Hung, Professor, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hung YC, Chen WC, Chang TC, Zheng HX, Liu YW, Tan YF, Lin SK, Lu YH, Hu WL, Tsai TM. Meridian study on the response current affected by electrical pulse and acupuncture. Nanoscale Res Lett. 2020 Jul 10;15(1):146. doi: 10.1186/s11671-020-03373-2. PMID 32651748
- [Background] Ifrim Chen F, Antochi AD, Barbilian AG. Acupuncture and the retrospect of its modern research. Rom J Morphol Embryol. 2019;60(2):411-418. PMID 31658313
- [Background] Zhang WB, Wang GJ, Fuxe K. Classic and Modern Meridian Studies: A Review of Low Hydraulic Resistance Channels along Meridians and Their Relevance for Therapeutic Effects in Traditional Chinese Medicine. Evid Based Complement Alternat Med. 2015;2015:410979. doi: 10.1155/2015/410979. Epub 2015 Mar 2. PMID 25821487
- [Derived] Lin CH, Tan YF, Tseng ST, Chen WC, Kuo CW, Wu CC, Tsai TM, Hu WL, Chang TC, Hung YC. Meridian study on the response current affected by acupuncture needling direction. Medicine (Baltimore). 2022 Sep 2;101(35):e30338. doi: 10.1097/MD.0000000000030338. PMID 36107585